CLINICAL TRIAL: NCT00921895
Title: A Comparison of the Sensitivity and Specificity of the RPS Adeno Detector IV™ at Detecting the Presence of Adenovirus to Viral Cell Culture.
Brief Title: A Comparison of the RPS Adeno Detector IV to Viral Cell Culture at Detecting Adenoviral Conjunctivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rapid Pathogen Screening (Industry)
Responsible Party: Sponsor
Organization: Lumos Diagnostics (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 200-003; NCT00799318 (obsolete NCT alias)
Record Dates: First submitted 2009-06-14; First posted 2009-06-16 (Estimated); Results first posted 2012-08-24 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Conjunctivitis
Keywords: Pink Eye,; Viral conjunctivitis; Adenoviral conjunctivitis; Keratoconjunctivitis
MeSH Terms: conditions — Conjunctivitis; Conjunctivitis, Viral; Keratoconjunctivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device Testing (Experimental): Patients with conjunctivitis will be tested with the RPS Adeno Detector IV
  Interventions: Device: RPS Adeno Detector IV

INTERVENTIONS:
Device: RPS Adeno Detector IV — One time test with the RPS Adeno Detector IV

SUMMARY:
To engage in a multi-center, prospective, masked clinical trial to investigate a non-invasive, rapid diagnostic test, the RPS Adeno Detector IV's ability to detect the presence of the adenovirus (ADV) antigen in cases of acute conjunctivitis by comparing it to cell culture with confirmatory immunofluorescence (CC-IFA). The polymerase chain reaction (PCR) will be used as a referee for discrepant cases.

DETAILED DESCRIPTION:
The RPS Adeno Detector IV will show substantial equivalence to cell culture for diagnosing adenoviral conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* A total of 150 patients will be enrolled and who present prospectively to either a private practice or academic center with a presumed diagnosis of acute viral conjunctivitis while an internal review board (IRB) approved ophthalmologist is available and determined by the ophthalmologist to have met the following criteria for the clinical diagnosis of acute viral conjunctivitis will be included in the study.
* Criteria for clinical diagnosis of viral conjunctivitis. Requires that patients are at least 1 month old and present within 7 days of developing a red eye with at least 1 criteria from each of the 3 categories below:

I History: 1) Spread from 1 eye to the other several days later, 2) a recent history of an upper respiratory infection (URI)

II Signs: 1) presence of follicles, 2) presence of a preauricular node

III Symptoms: 1) watery - purulent discharge, 2) eyelash matting, 3) itching, or 4) foreign body sensation

Exclusion Criteria:

* Patients with allergy to corn starch, talcum powder, or dacron will be excluded.
* Patients with a corneal ulcer or history of recent trauma will also be excluded.
* Any patients who are using any topical ointment (including OTC artificial tear ointments) in the last 72 hours should be excluded.
* Patients using other topical ophthalmic medications (i.e. antibiotics) must allow 60 minutes prior to device application following any topical ophthalmic drops.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shachar Tauber, MD, Principal Investigator — St John's Clinic; Jodi Luchs, MD, Principal Investigator — South Shore Eye Clinic; William Trattler, MD, Principal Investigator — Center For Excellence In Eye Care; Thomas Boland, MD, Principal Investigator — Northeastern Eye Institute; Michael DellaVecchia, MD/PhD, Principal Investigator — Wills Eye Institute; Murray Friedberg, MD, Principal Investigator — Manatee Eye Clinic; Chris Starr, MD, Principal Investigator — Weill Medical College of Cornell University; Marguerite McDonald, MD, Principal Investigator — Ophthalmic Consultants of Long Island
Locations (8):
- United States (8):
  - Manatee Eye Clinic, Bradenton, Florida
  - Center For Excellence in Eye Care, Miami, Florida
  - St John's Clinic, Springfield, Missouri
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - Weill-Cornell Medical College, New York, New York
  - South Shore Eye Care, Wantagh, New York
  - Wills Eye Institute, Philadelphia, Pennsylvania
  - Northeastern Eye Institute, Scranton, Pennsylvania

REFERENCES:
- [Derived] Sambursky R, Trattler W, Tauber S, Starr C, Friedberg M, Boland T, McDonald M, DellaVecchia M, Luchs J. Sensitivity and specificity of the AdenoPlus test for diagnosing adenoviral conjunctivitis. JAMA Ophthalmol. 2013 Jan;131(1):17-22. doi: 10.1001/2013.jamaophthalmol.513. PMID 23307204

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was June 2009 - May 2011. The study was performed at private ophthalmology practices and academic centers.
Period: Overall Study
Arm/Group | Device Testing
Started | 128
Completed | 128
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Device Testing
Number analyzed (Participants) | 128
Age, Customized [Median (Full Range); unit: years] | 43 [5 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 52
Region of Enrollment [Number; unit: participants]
  United States | 128

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of RPS Adeno Detector IV Compared to Cell Culture.
Description: Sensitivity is proportion of true positive cases compared to cell culture. Specificity is the proportion of true negative cases compared to cell culture.
Time Frame: 15 minutes
Measure: Number (95% Confidence Interval); unit: percentage of cases
Groups:
- RPS Adeno Detector IV (Sensitivity): Looking for the number of true positives as compared to cell culture.
- RPS Adeno Detector IV (Specificity): Looking for the number of true negatives as compared to cell culture.
Arm/Group | RPS Adeno Detector IV (Sensitivity) | RPS Adeno Detector IV (Specificity)
Number analyzed (Participants) | 31 | 97
percentage of cases | 90 [74.2 to 98.0] | 96 [89.8 to 98.9]

ADVERSE EVENTS:
Arm/Group | Device Testing
Serious Adverse Events (participants affected / at risk) | 0/128
Other Adverse Events (participants affected / at risk) | 0/128

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results to be published or presented shall be submitted to RPS for review and comment at least 30 days prior to submission for publication or presentation. Institution and/or PI may publish or present the results and data from the Institution's site individually (i) 12 months after conclusion, abandonment or termination of study at all sites, or (ii) after RPS confirms there will be no multicenter study publication, whichever occurs first.